CLINICAL TRIAL: NCT01459393
Title: Evaluation of the Formulation of 5-aminolevulinic Acid With Dimethylsulfoxide in Photodynamic Therapy for Treatment of Actinic Keratosis
Brief Title: Comparison Between 5-aminolevulinic Acid Photodynamic Therapy Versus Cryotherapy for Actinic Keratosis Treatment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Barretos Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5-ALAAK
Record Dates: First submitted 2011-10-12; First posted 2011-10-25 (Estimated); Last update posted 2017-06-28 (Actual); Status verified 2014-02

CONDITIONS: Actinic Keratosis
Keywords: Actinic keratosis; Photodynamic therapy; 5-aminolevulinic acid; Cryotherapy
MeSH Terms: conditions — Keratosis, Actinic | interventions — Cryotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 5-ALA Photodynamic Therapy (Experimental): Topical application of a 2mm of thickness layer of 20% 5-aminolevulinic acid (5-ALA) associated with 20% dimethyl sulfoxide (DMSO) and 3% ethylene diamine acid (EDTA) emulsion, over the actinic keratosis lesion and over a 0,5 cm margin around it. After a 4 hours interval under light protection with plastic film and aluminum foil, the light protection and the emulsion is removed. Then the lesion is lightened with a red (630 nm) incoherent LED lamp AKTILITE CL 128 (PhotoCure ASA, Oslo, Norway) with a total light dose of 37J/cm2.After that dressings are done and kept for 24H, and removed at patient home.
  Interventions: Drug: 5-ALA Photodynamic Therapy
- Cryotherapy with liquid nitrogen (Active Comparator): Topical application of liquid nitrogen spray (500ml Cry-ac ® bottle) over the actinic keratosis lesion and over a 0,5 cm margin around it during sufficient time to freeze both the lesion and margin.
  Interventions: Drug: Cryotherapy with liquid nitrogen

INTERVENTIONS:
Drug: 5-ALA Photodynamic Therapy
  Other Names: AKTILITE CL 128 (PhotoCure ASA, Oslo, Norway)
  Arms: 5-ALA Photodynamic Therapy
Drug: Cryotherapy with liquid nitrogen — Topical application of liquid nitrogen spray (500ml Cry-ac ® bottle) over the actinic keratosis lesion and over a 0,5 cm margin around it during sufficient time to freeze both the lesion and margin.
  Other Names: Cry-ac ®
  Arms: Cryotherapy with liquid nitrogen

SUMMARY:
This study aims to compare in a prospective and randomized way actinic keratosis treatment with 5-aminolevulinic acid photodynamic therapy versus cryotherapy, from the standpoint of therapeutic efficacy, pain, and cosmetic results.

DETAILED DESCRIPTION:
Actinic keratosis is a skin lesion induced by chronic sun exposure with a significant prevalence and malignant potential for squamous cell carcinoma, which makes essential its treatment. Today there are several possible therapies, where cryotherapy is usually applied in our practice. Photodynamic therapy (PDT)is another method also widespread for keratosis which involves the administration of a topical precursor drug which produces endogenous photosensitising substances activated by specific light, selectively destroying the diseased tissue. This study aims to evaluate the use the drug formulation for photodynamic therapy 5-aminolevulinic acid (5-ALA) associated with dimethyl sulfoxide, comparing its efficacy with conventional cryotherapy, and also pain and cosmetic results. This project enrolled 137 outpatients from the Department of Cutaneous Oncology of Barretos Cancer Hospital - Pio XII Foundation, with symmetrical and comparable keratosis in their upper limbs. With the same patient as controls, side arm and therapy to be used were randomized: cryotherapy or photodynamic therapy. For cryotherapy was utilized bottles of liquid nitrogen (Cry-ac, 500ml); and for photodynamic therapy was utilized incoherent red light lamp with a total dosis of 37J/cm² . There was one or two sessions of each therapy , at 0 and 3 months; and three assessments for evaluation were done at 0, 3 and 6 months of onset. The evaluations on efficacy were in terms of area regression, and classified as complete response or no response. Pain was assessed by visual analogue scale, and numerical scale. Cosmesis was evaluated with the presence or not, objectively, of hyper, hypopigmentation or scar retraction. Finally, patient's preference regarding utilized therapeutics was noted by the researcher.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years.
* Patients with actinic keratoses "symmetrical", ie, comparable in the upper limbs ( with the same grade, I, II or III).
* Patients in accordance with informed consent.

Exclusion Criteria:

* Patients with concomitant skin diseases, congenital or acquired (albinism, vitiligo, xeroderma, Gorlin, etc.)
* Immunosuppression (HIV, transplanted patients, etc.)
* Pregnancy or lactation
* Patients who do not agree with the informed consent initially or during the protocol.
* Presence of pigmented lesions near the keratoses.
* Patients with porphyria.
* Patients who have undergone less than 2 months with some kind of treatment for keratosis in the upper limbs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2010-11; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Complete response rates | 0 months (baseline), 3 months and 6 months
  Clinical evaluation of treated area.

SECONDARY OUTCOMES:
Visual Analogic Scale Pain Score | 0 months (baseline), 3 months, 6 months
  Pain was evaluated with a Visual Analogic Scale (blind) and a graduated scale. It was evaluated at the time 0 and 15 minutes after each intervention (Cryotherapy or PDT): at the first intervention (0 months), and at the second intervention if the residual lesion that indicates a second session (3 months).
  And at the third interwiew (6 months) there was no intervention, but the patients who was submitted to 2 interventions were requested about what intervention was more painfull (the first or the second one).
Cosmesis analysis | 3 months, 6 months
  Cosmesis was evaluated subjetively by the patient as one of the possibilities: aesthetic outcome awfull, bad, regular, good, excellent.
  Cosmesis was evaluated subjetively also by the researcher as one of the possibilities: aesthetic outcome awfull, bad, regular, good, excellent.
  And there was and objective evaluation of cosmesis by the researcher, the presece or absence of one or more of these criteria: hypochromia, hyperpigmentation,hyperemia, scar.

CONTACTS AND LOCATIONS:
Overall Officials: Catarina Robert, MD, Principal Investigator — Fundação Pio XII - Hospital de Câncer de Barretos; René AC Vieira, PHD, Study Director — Fundação Pio XII - Hospital de Câncer de Barretos; André L Carvalho, PHD, Study Director — Fundação Pio XII - Hospital de Câncer de Barretos
Locations (1):
- Barretos Cancer Hospital, Barretos, São Paulo, Brazil

REFERENCES:
- [Background] Braathen LR, Szeimies RM, Basset-Seguin N, Bissonnette R, Foley P, Pariser D, Roelandts R, Wennberg AM, Morton CA; International Society for Photodynamic Therapy in Dermatology. Guidelines on the use of photodynamic therapy for nonmelanoma skin cancer: an international consensus. International Society for Photodynamic Therapy in Dermatology, 2005. J Am Acad Dermatol. 2007 Jan;56(1):125-43. doi: 10.1016/j.jaad.2006.06.006. PMID 17190630
- [Background] De Rosa FS, Bentley MV. Photodynamic therapy of skin cancers: sensitizers, clinical studies and future directives. Pharm Res. 2000 Dec;17(12):1447-55. doi: 10.1023/a:1007612905378. PMID 11303952
- [Background] Dougherty TJ. A brief history of clinical photodynamic therapy development at Roswell Park Cancer Institute. J Clin Laser Med Surg. 1996 Oct;14(5):219-21. doi: 10.1089/clm.1996.14.219. No abstract available. PMID 9612186
- [Background] Fink-Puches R, Hofer A, Smolle J, Kerl H, Wolf P. Primary clinical response and long-term follow-up of solar keratoses treated with topically applied 5-aminolevulinic acid and irradiation by different wave bands of light. J Photochem Photobiol B. 1997 Nov;41(1-2):145-51. doi: 10.1016/s1011-1344(97)00096-1. PMID 9440322
- [Background] Fitzpatrick TB. The validity and practicality of sun-reactive skin types I through VI. Arch Dermatol. 1988 Jun;124(6):869-71. doi: 10.1001/archderm.124.6.869. No abstract available. PMID 3377516
- [Background] Freeman M, Vinciullo C, Francis D, Spelman L, Nguyen R, Fergin P, Thai KE, Murrell D, Weightman W, Anderson C, Reid C, Watson A, Foley P. A comparison of photodynamic therapy using topical methyl aminolevulinate (Metvix) with single cycle cryotherapy in patients with actinic keratosis: a prospective, randomized study. J Dermatolog Treat. 2003 Jun;14(2):99-106. doi: 10.1080/09546630310012118. PMID 12775317
- [Background] Glogau RG. The risk of progression to invasive disease. J Am Acad Dermatol. 2000 Jan;42(1 Pt 2):23-4. doi: 10.1067/mjd.2000.103339. PMID 10607353
- [Background] Jeffes EW, McCullough JL, Weinstein GD, Fergin PE, Nelson JS, Shull TF, Simpson KR, Bukaty LM, Hoffman WL, Fong NL. Photodynamic therapy of actinic keratosis with topical 5-aminolevulinic acid. A pilot dose-ranging study. Arch Dermatol. 1997 Jun;133(6):727-32. PMID 9197826
- [Background] Kaufmann R, Spelman L, Weightman W, Reifenberger J, Szeimies RM, Verhaeghe E, Kerrouche N, Sorba V, Villemagne H, Rhodes LE. Multicentre intraindividual randomized trial of topical methyl aminolaevulinate-photodynamic therapy vs. cryotherapy for multiple actinic keratoses on the extremities. Br J Dermatol. 2008 May;158(5):994-9. doi: 10.1111/j.1365-2133.2008.08488.x. Epub 2008 Mar 13. PMID 18341663
- [Background] Kennedy JC, Pottier RH. Endogenous protoporphyrin IX, a clinically useful photosensitizer for photodynamic therapy. J Photochem Photobiol B. 1992 Jul 30;14(4):275-92. doi: 10.1016/1011-1344(92)85108-7. PMID 1403373
- [Background] Malik Z, Kostenich G, Roitman L, Ehrenberg B, Orenstein A. Topical application of 5-aminolevulinic acid, DMSO and EDTA: protoporphyrin IX accumulation in skin and tumours of mice. J Photochem Photobiol B. 1995 Jun;28(3):213-8. doi: 10.1016/1011-1344(95)07117-k. PMID 7623186
- [Background] Moloney FJ, Collins P. Randomized, double-blind, prospective study to compare topical 5-aminolaevulinic acid methylester with topical 5-aminolaevulinic acid photodynamic therapy for extensive scalp actinic keratosis. Br J Dermatol. 2007 Jul;157(1):87-91. doi: 10.1111/j.1365-2133.2007.07946.x. Epub 2007 May 14. PMID 17501954
- [Background] Salasche SJ. Epidemiology of actinic keratoses and squamous cell carcinoma. J Am Acad Dermatol. 2000 Jan;42(1 Pt 2):4-7. doi: 10.1067/mjd.2000.103342. PMID 10607349
- [Background] Sotiriou E, Apalla Z, Maliamani F, Zaparas N, Panagiotidou D, Ioannides D. Intraindividual, right-left comparison of topical 5-aminolevulinic acid photodynamic therapy vs. 5% imiquimod cream for actinic keratoses on the upper extremities. J Eur Acad Dermatol Venereol. 2009 Sep;23(9):1061-5. doi: 10.1111/j.1468-3083.2009.03259.x. Epub 2009 Apr 8. PMID 19470041
- [Background] Szeimies RM, Karrer S, Radakovic-Fijan S, Tanew A, Calzavara-Pinton PG, Zane C, Sidoroff A, Hempel M, Ulrich J, Proebstle T, Meffert H, Mulder M, Salomon D, Dittmar HC, Bauer JW, Kernland K, Braathen L. Photodynamic therapy using topical methyl 5-aminolevulinate compared with cryotherapy for actinic keratosis: A prospective, randomized study. J Am Acad Dermatol. 2002 Aug;47(2):258-62. PMID 12140473
- [Background] Tschen EH, Wong DS, Pariser DM, Dunlap FE, Houlihan A, Ferdon MB; Phase IV ALA-PDT Actinic Keratosis Study Group. Photodynamic therapy using aminolaevulinic acid for patients with nonhyperkeratotic actinic keratoses of the face and scalp: phase IV multicentre clinical trial with 12-month follow up. Br J Dermatol. 2006 Dec;155(6):1262-9. doi: 10.1111/j.1365-2133.2006.07520.x. PMID 17107399
- [Background] Yantsos VA, Conrad N, Zabawski E, Cockerell CJ. Incipient intraepidermal cutaneous squamous cell carcinoma: a proposal for reclassifying and grading solar (actinic) keratoses. Semin Cutan Med Surg. 1999 Mar;18(1):3-14. doi: 10.1016/s1085-5629(99)80003-0. PMID 10188837